CLINICAL TRIAL: NCT04703218
Title: REEDUCATION OF OLFACTORY DISORDERS AFTER A CEREBRAL VASCULAR ACCIDENT IN ADULTS
Acronym: RE-OLF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of patients
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-055
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Adult With Stroke and Olfaction's Complaint
MeSH Terms: interventions — Olfactory Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with stroke and olfaction disorder benefiting from specific olfaction training. (Experimental)
  Interventions: Other: olfactory rehabilitation
- Patients with stroke and olfactory disorder benefiting from standard post-stroke rehabilitation (No Intervention)

INTERVENTIONS:
Other: olfactory rehabilitation — Olfactory rehabilitation consists of smelling 4 scents twice a day using scent sticks, for 12 weeks
  Arms: Patients with stroke and olfaction disorder benefiting from specific olfaction training.

SUMMARY:
Study context:

The literature identifies more and more research revealing olfactory disorders, with a high frequency after an acquired brain injury. So far, studies have mainly focused on post-traumatic and post-infectious olfactory disorders of the upper airways. There is scarcer data available on the olfactory disorders occurring after stroke. A recent study found 43.6% of patients with a loss of olfactory function after a stroke (2). This type of disorder can have repercussions in everyday life and endanger people, not being able to smell a burning odor or gas fumes. In addition, patients frequently describe loss of pleasure associated with these olfactory disorders (3). Tests allowing the evaluation of these difficulties exist but remain little used in clinical routine (4). These psychophysical tests allow a quantitative analysis of the olfactory capacities of subjects through various measures such as the detection threshold (T SST sub-score), discrimination (D SST sub-score) or the identification of an odor. (SST sub-score I). Some studies have shown a reduction in olfactory disturbances following specific training. Thus, Hummel et al. proposed a self-stimulation protocol to patients whose olfactory dysfunction was due to various aetiologies (post-infectious, post-traumatic or idiopathic) (5). People were to smell 4 scents twice a day for 12 weeks. The results show an improvement in the olfaction of the patients, while no change was noted in the subjects who did not perform the training. Lehrer et al. obtained similar results in patients with head trauma (CT) after 3 months of training (6). However, no study has looked at the effect of specific olfaction training in post-stroke patients. The few data available in the literature suggest that these disorders are common after stroke.

Objectives :

We propose an open, randomized controlled study, comparing the SST score between the group of patients who received olfactory training and the group who received standard rehabilitation.

Material and methods :

In the treatment of post-stroke olfactory disorders, we will suggest to patients hospitalized in SSR or followed in consultation to participate in a controlled, randomized open study.

All included patients will be assessed using the SST and the modified ASOF quality of life questionnaire (7). After randomization, patients in the treatment group will benefit from a presentation of specific olfaction training. This training consists of smelling 4 scents twice a day using scent sticks, for 12 weeks. At the end of these 12 weeks, a post-protocol evaluation including the SST, the modified ASOF quality of life questionnaire and a measurement of any side effects related to training will be offered.

Hypothesis tested:

The aim of this work is to evaluate the effectiveness of a specific olfaction training protocol in patients with olfaction disorders following stroke.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient under 65 in order to avoid presbyosmia bias,
* Patient suffering from an ischemic and / or hemorrhagic stroke dating at least 3 months,
* Patient followed in the SRH department and / or in post-stroke consultation,
* French-speaking patient,
* Patient affiliated to the social security scheme,
* Patient having signed the informed consent.

Exclusion Criteria:

* Patient with a TDI score greater than 30.5 on the SST,
* Patient with global aphasia: score <25 on the oral comprehension subtest of MT86 sentences (1),
* Person under legal protection (guardianship, curatorship, safeguard of justice),
* Patient treated with corticosteroids, corticosteroids, steroids, antihistamines and antibiotics which may have repercussions on olfaction,
* History of trauma to the face,
* History of ENT surgery,
* Chronic rhinitis,
* Infection of the ENT sphere in the 15 days preceding inclusion,
* Neurodegenerative pathology,
* Parosmia, phantosmia or cacosmia,
* History of systemic chemotherapy or radiotherapy to the head.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
TDI score obtained in SST after the training period (12 weeks) | 3 months

SECONDARY OUTCOMES:
Score obtained on the ASOF quality of life questionnaire modified after training (12 weeks) | 3 months
T, D and I sub-scores obtained in SST after training (12 weeks) | 3 months
Number of complaints about side effects and possible discomfort related to training | 3 months and 6 months
Number of training stops (training < 12 weeks) | 3 months
score obtained in the SST after training (12 weeks) | 3 months
TDI score obtained at SST 3 months after the end of training (at 24 weeks) | 6 months
Percentage of patients changing category according to the thresholds validated by the SST (anosmia, hyposmia, normosmia). | 3 months and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No